CLINICAL TRIAL: NCT00168337
Title: A Study of the Safety and Efficacy of a New Treatment for Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206207-011
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone 700 μg (Experimental): 700 µg Dexamethasone posterior segment drug delivery system - injection into the vitreous cavity not less than every 6 months for up to 36 months.
  Interventions: Drug: Dexamethasone
- Dexamethasone 350 μg (Experimental): 350 µg Dexamethasone posterior segment drug delivery system - injection into the vitreous cavity not less than every 6 months for up to 36 months.
  Interventions: Drug: Dexamethasone
- Sham (Sham Comparator): Sham posterior segment drug delivery system - needle-less drug delivery system without study medication not less than every 6 months for up to 36 months.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Dexamethasone — 350 µg or 700 µg dexamethasone posterior segment drug delivery system - injection into the vitreous cavity not less than every 6 months for up to 36 months.
  Other Names: Posurdex®; Ozurdex®
  Arms: Dexamethasone 350 μg; Dexamethasone 700 μg
Other: Sham — Sham posterior segment drug delivery system-needle-less drug delivery system without study medication not less than every 6 months for up to 36 months.
  Arms: Sham

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal implant of dexamethasone for the treatment of diabetic macular edema.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older with diabetic macular edema;
* Decrease in visual acuity in at least one eye as a result of macular edema (20/50 or worse);
* Visual acuity in other eye no worse than 20/200

Key Exclusion Criteria:

* Known anticipated need for ocular surgery within next 12 months;
* History of glaucoma or current high eye pressure requiring more than 1 medication;
* Uncontrolled systemic disease;
* Known steroid-responder;
* Use of systemic steroids;
* Use of Warfarin/Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2005-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (14):
- Artesia, California, United States
- São Paulo, Brazil
- Mississauga, Ontario, Canada
- Bogotá, Colombia
- Dijon, France
- Budapest, Hungary
- New Delhi, India
- Milan, Italy
- Auckland, New Zealand
- Warsaw, Poland
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan
- London, United Kingdom

REFERENCES:
- [Derived] Blinder KJ, Wykoff CC, Ferencz JR, Ehlers JP, Fang Y, Lai H, Ogidigben M, Lopez FJ. IMPACT OF THE DEXAMETHASONE IMPLANT ON SLOWING DIABETIC RETINOPATHY PROGRESSION: Post Hoc Analysis of the MEAD Study. Retina. 2025 Dec 1;45(12):2252-2262. doi: 10.1097/IAE.0000000000004623. PMID 40712145
- [Derived] Kozak I, Do DV, Lai H, Ogidigben MJ, Lopez FJ. Time-in-Range Analysis of Responses after Intravitreal Dexamethasone Therapy in Eyes with Diabetic Macular Edema. Ophthalmol Sci. 2025 May 26;5(5):100833. doi: 10.1016/j.xops.2025.100833. eCollection 2025 Sep-Oct. PMID 40688490
- [Derived] Valentim CCS, Lai H, Ogidigben MJ, Singh RP, Talcott KE. Baseline factors affecting diabetic macular oedema resolution after intravitreal dexamethasone implant treatment: post hoc analysis of the MEAD study. BMC Ophthalmol. 2025 Jul 9;25(1):403. doi: 10.1186/s12886-025-04208-3. PMID 40634898
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Yoon YH, Boyer DS, Maturi RK, Bandello F, Belfort R Jr, Augustin AJ, Li XY, Bai Z, Hashad Y; Ozurdex MEAD Study Group. Natural history of diabetic macular edema and factors predicting outcomes in sham-treated patients (MEAD study). Graefes Arch Clin Exp Ophthalmol. 2019 Dec;257(12):2639-2653. doi: 10.1007/s00417-019-04464-2. Epub 2019 Oct 25. PMID 31654188
- [Derived] Danis RP, Sadda S, Li XY, Cui H, Hashad Y, Whitcup SM. Anatomical effects of dexamethasone intravitreal implant in diabetic macular oedema: a pooled analysis of 3-year phase III trials. Br J Ophthalmol. 2016 Jun;100(6):796-801. doi: 10.1136/bjophthalmol-2015-306823. Epub 2015 Nov 18. PMID 26581718
- [Derived] Augustin AJ, Kuppermann BD, Lanzetta P, Loewenstein A, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Dexamethasone intravitreal implant in previously treated patients with diabetic macular edema: subgroup analysis of the MEAD study. BMC Ophthalmol. 2015 Oct 30;15:150. doi: 10.1186/s12886-015-0148-2. PMID 26519345

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Started | 188 | 181 | 185
Completed | 118 | 112 | 82
Not Completed | 70 | 69 | 103

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham | Total
Number analyzed (Participants) | 188 | 181 | 185 | 554
Age, Customized [Number; unit: Participants]
  <45 years | 2 | 8 | 6 | 16
  45 to 65 years | 116 | 109 | 108 | 333
  >65 years | 70 | 64 | 71 | 205
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 75 | 70 | 222
  Male | 111 | 106 | 115 | 332

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Best Corrected Visual Acuity (BCVA) Improvement of ≥15 Letters From Baseline in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates improvement and a decrease in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 188 | 181 | 185
Percentage of Patients | 22.3 | 18.2 | 10.8

2. Secondary Outcome: Average Change From Baseline in BCVA in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The average BCVA is calculated across study visits for each patient. A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, 39 Months
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 188 | 181 | 185
Letters
  Baseline | 55.9 (9.83) | 55.2 (9.69) | 57.0 (8.76)
  Average Change from Baseline Over 39 months | 2.9 (8.55) | 2.9 (7.67) | 2.0 (8.20)

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 188 | 181 | 185
Letters
  Baseline | 55.9 (9.83) | 55.2 (9.69) | 57.0 (8.76)
  Change from Baseline at Month 39/Final Visit | 1.3 (17.03) | 1.4 (15.17) | -0.0 (15.41)

4. Secondary Outcome: Percentage of Patients With a BCVA Improvement of ≥10 Letters From Baseline in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 188 | 181 | 185
Percentage of Patients | 34.6 | 29.8 | 24.9

5. Secondary Outcome: Change From Baseline in Retinal Thickness as Measured by Optical Coherence Tomography (OCT)
Description: OCT is a laser-based, noninvasive, diagnostic system that provides high-resolution, three-dimensional images of the retina from which retinal thickness can be measured. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 186 | 179 | 177
Microns
  Baseline | 486.0 (163.12) | 475.4 (160.70) | 453.7 (135.36)
  Change from Baseline at Month 39/Final Visit | -117.9 (227.16) | -131.2 (204.33) | -70.4 (180.82)

6. Post Hoc Outcome: 10th Percentile for Time to BCVA Improvement of ≥15 Letters From Baseline in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). Shorter durations of time to improvement are best. The 10th percentile represents the first 10% of patients to reach a BCVA improvement of ≥15 letters from baseline in the study eye.
Time Frame: Baseline, 39 Months
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Days
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 188 | 181 | 185
Days | 50 [24 to NA] | 49 [33 to NA] | 186 [33 to NA]

7. Post Hoc Outcome: Percentage of Patients With BCVA Improvement of ≥15 Letters From Baseline in the Study Eye at 3-month Intervals
Description: as for outcome 1
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, Month 24, Month 27, Month 30, Month 33, Month 36, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 188 | 181 | 185
Percentage of Patients
  Month 3 | 11.7 | 14.4 | 2.7
  Month 6 | 8.5 | 6.1 | 3.2
  Month 9 | 15.4 | 14.4 | 7.0
  Month 12 | 12.8 | 9.9 | 9.7
  Month 15 | 12.8 | 14.4 | 9.7
  Month 18 | 12.2 | 10.5 | 9.2
  Month 21 | 15.4 | 9.4 | 10.3
  Month 24 | 18.1 | 9.4 | 10.3
  Month 27 | 16.5 | 12.2 | 10.3
  Month 30 | 18.6 | 12.2 | 10.3
  Month 33 | 18.6 | 14.4 | 9.7
  Month 36 | 19.7 | 16.6 | 10.8
  Month 39/Final Visit | 22.3 | 18.2 | 10.8

ADVERSE EVENTS:
Description: The Safety Population included all treated patients and was used for adverse event (AE) and Serious Adverse Event (SAE) reporting.
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Serious Adverse Events (participants affected / at risk) | 63/187 | 68/178 | 49/186
Other Adverse Events (participants affected / at risk) | 180/187 | 172/178 | 157/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dexamethasone 700 μg (N=187) | Dexamethasone 350 μg (N=178) | Sham (N=186)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia of Chronic Disease (Blood and lymphatic system disorders) | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 3 | 3 | 1
Acute Coronary Syndrome (Cardiac disorders) | 2 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 6 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 4 | 2
Angina Unstable (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac Disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Insufficiency (Cardiac disorders) | 0 | 1 | 0
Pulseless Electrical Activity (Cardiac disorders) | 0 | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 8 | 7 | 2
Vitreous Haemorrhage (Eye disorders) | 8 | 2 | 4
Macular Oedema (Eye disorders) | 2 | 3 | 0
Macular Fibrosis (Eye disorders) | 2 | 1 | 2
Retinal Detachment (Eye disorders) | 2 | 0 | 0
Cataract Subcapsular (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Necrotising Retinitis (Eye disorders) | 1 | 0 | 0
Open Angle Glaucoma (Eye disorders) | 1 | 0 | 0
Cataract Cortical (Eye disorders) | 0 | 1 | 0
Cystoid Macular Oedema (Eye disorders) | 0 | 1 | 0
Diabetic Retinal Oedema (Eye disorders) | 0 | 0 | 1
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 1
Hyalosis Asteroid (Eye disorders) | 0 | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Pelvic Mass (General disorders) | 1 | 0 | 0
Medical Device Complication (General disorders) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Device Dislocation (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 3 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 0
Endophthalmitis (Infections and infestations) | 2 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Incision Site Infection (Infections and infestations) | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Pneumonia Viral (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 1
Gallbladder Empyema (Infections and infestations) | 0 | 0 | 1
Localised Infection (Infections and infestations) | 0 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Comminuted Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Meniscal Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Eagles Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/111 | 3/106 | 1/115
Benign Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Squamous Cell Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/77 | 0/75 | 0/70
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 2 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 2 | 3
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0 | 1
Altered State of Consciousness (Nervous system disorders) | 1 | 0 | 0
Benign Intracranial Hypertension (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0
VIIth Nerve Paralysis (Nervous system disorders) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1
Cervical Myelopathy (Nervous system disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 2 | 2
Renal Failure (Renal and urinary disorders) | 1 | 1 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 2 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1 | 3
Calculus Ureteric (Renal and urinary disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1/111 | 1/106 | 0/115
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1/111 | 0/106 | 0/115
Uterine Haemorrhage (Reproductive system and breast disorders) | 1/77 | 0/75 | 0/70
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Victim of Homicide (Social circumstances) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Malignant Hypertension (Vascular disorders) | 1 | 0 | 0
Extremity Necrosis (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 1 | 0
Temporal Arteritis (Vascular disorders) | 0 | 1 | 0
Venous Insufficiency (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 700 μg (N=187) | Dexamethasone 350 μg (N=178) | Sham (N=186)
Cataract (Eye disorders) | 78 | 65 | 29
Intraocular Pressure Increased (Investigations) | 50 | 51 | 15
Conjunctival Haemorrhage (Eye disorders) | 39 | 40 | 28
Hypertension (Vascular disorders) | 35 | 31 | 15
Macular Oedema (Eye disorders) | 30 | 27 | 20
Visual Acuity Reduced (Eye disorders) | 27 | 30 | 12
Cataract Subcapsular (Eye disorders) | 25 | 22 | 8
Diabetic Retinal Oedema (Eye disorders) | 24 | 23 | 18
Vitreous Haemorrhage (Eye disorders) | 22 | 32 | 26
Macular Fibrosis (Eye disorders) | 21 | 29 | 12
Ocular Hypertension (Eye disorders) | 19 | 13 | 6
Retinal Exudates (Eye disorders) | 16 | 12 | 12
Dry Eye (Eye disorders) | 15 | 10 | 7
Vitreous Detachment (Eye disorders) | 12 | 14 | 8
Lenticular Opacities (Eye disorders) | 12 | 6 | 3
Retinal Haemorrhage (Eye disorders) | 11 | 17 | 9
Urinary Tract Infection (Infections and infestations) | 11 | 8 | 9
Diabetic Retinopathy (Eye disorders) | 10 | 14 | 9
Conjunctival Oedema (Eye disorders) | 10 | 10 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 4 | 6
Conjunctival Hyperaemia (Eye disorders) | 9 | 12 | 11
Anaemia (Blood and lymphatic system disorders) | 9 | 10 | 8
Oedema Peripheral (General disorders) | 9 | 10 | 6
Blood Creatinine Increased (Investigations) | 9 | 9 | 8
Eye Pain (Eye disorders) | 8 | 13 | 10
Punctate Keratitis (Eye disorders) | 8 | 9 | 7
Retinal Neovascularisation (Eye disorders) | 6 | 16 | 14
Cataract Cortical (Eye disorders) | 6 | 11 | 9
Retinal Aneurysm (Eye disorders) | 6 | 9 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 13 | 7
Blepharitis (Eye disorders) | 4 | 3 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.